CLINICAL TRIAL: NCT04674683
Title: A Multicenter, Randomized, Double-Blind Phase 3 Study of HBI-8000 Combined With Nivolumab Versus Placebo With Nivolumab in Patients With Unresectable or Metastatic Melanoma Not Previously Treated With PD-1 or PD-L1 Inhibitors
Brief Title: Study Comparing Investigational Drug HBI-8000 + Nivolumab vs. Placebo + Nivolumab in Patients With Advanced Melanoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBI-8000-303
Record Dates: First submitted 2020-12-07; First posted 2020-12-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Unresectable or Metastatic Melanoma; Progressive Brain Metastasis
Keywords: HBI-8000; nivolumab; melanoma; brain metastasis
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — HBI-8000; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled Phase 3 study of HBI-8000 or Placebo combined with nivolumab.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All Eligible patients will be randomized within the appropriate stratum at a 1:1 ratio to the Test arm or the Control arm, with the exception of Cohort for special population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Arm (Experimental): HBI-8000 30 mg oral BIW + nivolumab IV at specific doses on specific days
  Interventions: Drug: HBI-8000 in combination with nivolumab
- Control Arm (Placebo Comparator): Placebo oral BIW + nivolumab IV at specific doses on specific days
  Interventions: Drug: Placebo in combination with nivolumab

INTERVENTIONS:
Drug: HBI-8000 in combination with nivolumab — Patients will take 30 mg of HBI-8000 orally approximately 30 minutes after a full meal, beginning on Day 1 and continue every 3 to 4 days on the BIW schedule. On Day 1 of each cycle nivolumab IV will be administered by intravenous infusion at specific doses on specific days in accordance with OPDIVO® manufacturer regional product information insert and the institution's prescribing practice. In adolescent patients with body weight < 40 kg, nivolumab will be dosed at specific doses on specific days.
  Other Names: For HBI-8000: tudicdinostat; For nivolumab: OPDIVO®
  Arms: Test Arm
Drug: Placebo in combination with nivolumab — Patients will take 30 mg of Placebo orally approximately 30 minutes after a full meal, beginning on Day 1 and continue every 3 to 4 days on the BIW schedule. On Day 1 of each cycle nivolumab IV at specific doses will be administered by intravenous infusion in accordance with OPDIVO® manufacturer regional product information insert and the institution's prescribing practice.
  Other Names: For nivolumab: OPDIVO®
  Arms: Control Arm

SUMMARY:
This is a clinical study to compare the efficacy and safety of HBI-8000 combined with nivolumab to Placebo combined with nivolumab in patients with unresectable or metastatic melanoma. A separate open-label cohort of adults with new, progressive brain metastasis or adolescents with or without new progressive brain metastasis receive HBI-8000 combined with nivolumab.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 3 study of HBI-8000 or Placebo combined with nivolumab. Randomization of eligible patients will be stratified by PD-L1 expression (positive, ≥1% expression level versus negative, <1% expression level) and LDH (normal versus elevated) in the main study. Adults with new, progressive brain metastasis, or adolescents with or without new progressive brain metastasis will be enrolled in a separate, non-randomized, open-label cohort to receive the combination of HBI-8000 and nivolumab.

In the main study, eligible patients will be randomized within the appropriate stratum at a 1:1 ratio to the Test arm or the Control arm. Study treatment will be initiated within 3 days of randomization.

A treatment cycle consists of 28 days. Patients will be treated with one of the following:

Test arm: HBI-8000 30 mg oral BIW + nivolumab IV at specific doses on specific days

Control arm: Placebo oral BIW + nivolumab IV at specific doses on specific days

The Study Treatment (HBI-8000 or Placebo) is administered approximately 30 minutes after a full meal.

The Study Treatment (HBI-8000 or Placebo) will be administered twice a week on the following days of every 28-day cycle:

* CxW1: Days 1, 4
* CxW2: Days 8, 11
* CxW3: Days 15, 18
* CxW4: Days 22, 25

Study treatment must commence within 3 days after randomization and continue up to 2 years or until disease progression (confirmed), unacceptable toxicity or patient withdrawal of consent.

In addition to Study Treatment, nivolumab is administered at specific doses on specific days as an intravenous infusion over approximately 30 minutes. Nivolumab will be administered on Day 1 of each cycle.

For non-randomized cohort for special population, eligible subjects will receive HBI-8000 30 mg oral BIW and nivolumab IV at specific doses on specific days, under the same schedule as described above. For adolescents weighing < 40 kg, nivolumab will be dosed at specific doses every 4 weeks. Nivolumab will be administered on Day 1 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed diagnosis of non-uveal, Stage III (unresectable), or Stage IV (metastatic) melanoma according to AJCC staging system (8th edition).
2. Known BRAF V600 mutation status or consent to BRAF V600 mutation testing before randomization.
3. Tumor tissue available for PD-L1 testing at central lab or local laboratory; results must be obtained prior to randomization. In the event when archived tumor tissue is not available, new tumor biopsy or historical PD-L1 test results may be used for randomization, however tumor tissue, either taken previously or newly acquired, must be provided for central biomarker confirmation for final data analyses.

   PD-L1 expression level is required for randomization. In order to be randomized, a patient must be classified as PD-L1 positive or PD-L1 negative according to the following criteria:
   * PD-L1 positive (≥ 1% tumor cell membrane staining in a minimum of a hundred evaluable tumor cells) vs
   * PD-L1 negative (< 1% tumor cell membrane staining in a minimum of a hundred evaluable tumor cells).

   Note: If an insufficient amount of tumor tissue is available prior to the start of the screening phase, patients must consent to allow the acquisition of additional tumor tissue for performance of biomarker analyses.
4. Males or females 12 years of age or older.
5. ECOG performance status ≤1 for age ≥18 years, Lansky performance status ≥80% for age 12 to 17 years.
6. At least one measurable lesion defined by RECIST 1.1 criteria, (separate from the lesion to be used for tumor tissue collection) not counting brain metastasis with:

   * Longest diameter ≥10 mm by CT (when slice thickness is ≤5 mm); or ≥ 2× slice thickness (when slice thickness is >5 mm)
   * Pathologically enlarged lymph node: ≥15 mm in short axis by CT (when slice thickness is ≤5 mm)
   * Clinical: ≥10 mm (that can be accurately measured with calipers).
7. Have not received anti-PD-1, anti-PD-L1 or other systemic therapy for unresectable or metastatic melanoma, except for the following, provided that the patient has recovered from all treatment-related toxicities:

   * BRAF mutation targeting therapy > 4 weeks before administration of Study Treatment.
   * Adjuvant or neoadjuvant therapy with PD-1 or PD-L1 inhibitors or anti-cytotoxic T lymphocyte-associated protein 4 (anti-CTLA-4) is allowed if disease progression/or recurrence had occurred at least 6 months after the last dose of neoadjuvant/adjuvant therapy and prior to receiving the first dose on this study and no clinically significant immune related toxicities leading to treatment discontinuation were observed
   * Adjuvant interferon therapy must have been completed > 6 weeks before administration of Study Treatment
8. Any prior radiotherapy or minor surgery must be completed at least 2 weeks and 1 week respectively before Day 1 dosing and recovered from all treatment related toxicities
9. Screening laboratory results within 14 days prior to randomization:

   * Hematology: WBC ≥3000/μL, neutrophils ≥1500/μL, platelets ≥100 × 103/μL, hemoglobin ≥10.0 g/dL independent of transfusion. The use of erythropoietic growth factor to achieve hemoglobin (Hgb) ≥ 10 g/dl is acceptable.
   * The CrCL≥ 30 mL/min using Cockcroft-Gault formula.
   * AST and ALT ≤3 × ULN, alkaline phosphatase ≤2.5 × ULN unless bone metastases present (patients with documented bone metastases: alkaline phosphatase <5 x ULN), bilirubin ≤ 1.5 × ULN (unless known Gilbert's disease where it must be ≤ 3 × ULN), serum albumin ≥ 3.0 g/dL).
10. Negative serum pregnancy test at baseline for women of childbearing potential.
11. Females of childbearing potential (non-surgically sterile or premenopausal female capable of becoming pregnant) and all males (due to potential risk of drug exposure through the ejaculate) must agree to use adequate birth control measures from study start, during the study and for 5 months after the last dose of Study Drug. Acceptable methods of birth control in this trial include two highly effective methods of birth control (as determined by the Investigator; one of the methods must be a barrier technique) or abstinence.
12. Have the ability to understand and the willingness to sign a written informed consent document, comply with study scheduled treatment, visits and assessments.

Exclusion Criteria:

1. History of ≥ Grade 3 hypersensitivity reactions to monoclonal antibodies.
2. Previous treatment with a PD-1, PD-L1, PD-L2, CTLA-4 inhibitor, or any other agents targeting T-cell co-stimulation or immune checkpoint pathways for unresectable or metastatic melanoma.
3. Recipient of solid organ transplant.
4. History of a cardiovascular illness including: congestive heart failure (New York Heart Association Grade III or IV); unstable angina or myocardial infarction within the previous 6 months prior to first dose of Study Treatment; or symptomatic cardiac arrhythmia despite medical management. QT interval corrected by heart rate using QTcF >450 ms in males or >470 ms in females, or congenital long QT syndrome.
5. Uncontrolled hypertension, systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100 mmHg.
6. Patients with new, active, or progressive brain metastases or leptomeningeal disease with except when considered for a separate special open-label cohort.
7. History of hemorrhagic diarrhea, inflammatory bowel disease, active uncontrolled peptic ulcer, or bowel resection that affects absorption of orally administered drugs.
8. Active, known, or suspected autoimmune disease, except for Type I diabetes mellitus, hypothyroidism requiring only hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic therapy.
9. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
10. Known history of testing positive for HIV, known AIDS.
11. Hepatitis B surface antigen positive or hepatitis C antibody positive. Further investigation per institutional practices may be performed to exclude active infection.
12. Patients with a condition requiring chronic systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days before administration of Study Treatment. Inhaled or topical steroids, or adrenal replacement dose of corticosteroids at dose ≤ 10 mg/day prednisone equivalent are permitted.
13. Use of another investigational agent (drug or vaccine not marketed for any indication) within 28 days or before administration of Study Treatment. If the investigational agent is a monoclonal antibody then within 3 months before administration of Study Treatment
14. Pregnant or breast-feeding women.
15. Have a history of any other malignancy unless in remission for 2 years or locally curable cancers that have been treated with curative intent with no evidence of recurrence, such as:

    * Basal or squamous cell skin cancer
    * Superficial bladder cancer
    * Carcinoma in situ of cervix or breast
    * Incidental prostate cancer
    * Non melanomatous skin cancer
    * Prostate cancer treated with curative intent with serum prostate specific antigen (PSA) < 2.0 ng/mL
16. Patients with medical conditions requiring administration of strong cytochrome P450 (CYP), CYP3A4 Inducers and Inhibitors with no alternative therapy.
17. Uncontrolled adrenal insufficiency or active chronic liver disease.
18. Has received approved live vaccine/live attenuated vaccines within 30 days of planned Cycle 1 Day 1. Inactivated viral vaccines or vaccines based upon subviral component are allowed; however intranasal influenza vaccines (e.g. Flu-Mist) are not allowed. COVID-19 vaccination should be administered at least 7 days before Cycle 1 Day 1.
19. Underlying medical conditions that, in the Investigator's opinion, will make the administration of Study Treatment hazardous or obscure the interpretation of toxicity determination or AEs.
20. Patients with a history of or active interstitial lung disease (ILD) or non-infectious pneumonitis.
21. Patients with prior organ or hematopoietic cell transplant (HCT), including allogeneic HCT.
22. Patients with known sensitivity to any of the ingredients of the Study Treatment.
23. Patients who received radiation therapy within 14 days of the first dose of the Study Treatment.
24. Patients who take drugs that prolong the QT interval or cause torsades de pointes or produce significant ventricular dysrhythmias.
25. Patients that are unwilling or unable to comply with procedures required in this protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | From date of randomization to the earliest date of documented progressive disease (PD), assessed up to 48 months
  Progression-free Survival (PFS) defined as the time (in days) from the date of randomization to the first date of documented disease progression as determined by BIRC, or the date of death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until disease progression or unacceptable toxicity, assessed up to 48 months
  Objective Response Rate (ORR) defined as the percentage of patients enrolled in each study arm with a best response of Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1), as determined by the blinded independent review committee (BIRC).
Overall Survival | From date of randomization to death due to any cause, assessed up to 48 months
  Overall Survival (OS) defined as the time from randomization date to the date of death due to any cause.
Safety, defined as the incidence rate of AEs | From date of screening until the end of study, assessed up to 48 months
  Safety, defined as the incidence rate of AEs. The NCI-CTCAE v5.0 will serve as the reference document for choosing the appropriate terminology to grade the severity of AEs, and to assess the causal relationship and outcomes.

OTHER OUTCOMES:
Duration of Response | Assessed up to 48 months
  Duration of Response (DoR), defined as the time from the first date of objective response (PR or CR) according to RECIST 1.1 as determined by the BIRC to the first date of progressive disease (PD) or death from any cause.
Disease Control Rate | Assessed up to 48 months
  Disease Control Rate (DCR), defined as the percentage of total patients enrolled in each study arm with a best response of CR, PR or SD according to RECIST 1.1, as determined by the BIRC.
Time to Response | Assessed up to 48 months
  Time to Response (TTR), defined as the time from the date of randomization to the first date of documented objective response (CR or PR) as determined by the BIRC.
Time to Progression | Assessed up to 48 months
  Time to Progression (TTP) defined as the time from the date of randomization to the first date of documented progression as determined by the BIRC. For patients with no PD, TTP will be considered censored at death or at the last evaluable imaging date.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Lee, MD, PhD, Study Director — HUYABIO International, LLC.
Locations (139):
- United States (31):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Innovative Clinical Research Institute (ICRI), Pasadena, California
  - Emad Ibrahim, MD, INC, Redlands, California
  - Kaiser Permanente Oncology Research, Riverside, California
  - California Cancer Associates for Research and Excellence, Inc. (cCARE), San Marcos, California
  - Boca Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Ascension Sacred Heart Medical Oncology, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Goshen Center for Cancer Care, Goshen, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Frederick Memorial Healthcare System, Frederick, Maryland
  - St Louis Cancer Care, Bridgeton, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - St. Vincent - Frontier Cancer Center, Billings, Montana
  - Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Thomas Jefferson University Medical Oncology Clinic, Philadelphia, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Carolina Blood and Cancer Care Associates, Lancaster, South Carolina
  - Renovatio Clinical, The Woodlands, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Froedtert Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (10):
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - University of the Sunshine Coast, Buderim, Queensland
  - Icon Cancer Centre Wesley, South Brisbane, Queensland
  - Ballarat Health Services, Ballarat, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Royal Brisband and Women's Hospital, Brisbane
  - Liverpool Hospital, Liverpool
  - Affinity Clinical Research, Nedlands
  - Tweed Hospital, Tweed Heads
  - Calvary Mater Newcastle, Waratah
- Austria (2):
  - Medical University of Graz Department of Dermatology and Venerology, Graz
  - Univ.-Lkinik für Dermatologie, Venerologie und Allergologie, Innsbruck
- Belgium (6):
  - AZ Klina, Brasschaat
  - Cliniques Universitaires, Brussels
  - AZ Maria Middelares, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Hospital de la Citadelle, Liège
  - Clinique Saint-Pierre, Ottignies
- Brazil (13):
  - Ensino e Terapia de Inovação Clίnica AMO-ETICA, Salvador, Estado de Bahia
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer,, Curitiba, Paraná
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital São Vicente de Paulo, Centro, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Centro Gaúcho Integrado de Oncologia, Hematologia, Porto Alegre, Rio Grande do Sul
  - Hospital de Clίnίcas de Porto Alegre, Santa Cruz do Sul, Rio Grande do Sul
  - Oncosite-Centro de Pesquisa Clίnica em Oncologia, São Cristóvão, Rio Grande do Sul
  - Hopital de Câncer de Barretos-Fundação Pio XII, Barretos, São Paulo
  - Fundação Doutor Amaral Carvalho, Jaú, São Paulo
  - CEPHO-Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de São Paulo - "Octavio Frias de Oliveira"-ICESP, São Paulo, São Paulo
- Czechia (3):
  - Fakultni nemocnice Olomoue, Olomouc
  - Fakultni nemocnice Ostrava Kozni oddeleni, Ostrava-Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- France (10):
  - CHU de Besançon - Hôpital Jean MINJOZ, Besançon
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Dijon, Service de dermatologie, Dijon
  - CHU Grenoble Alpes, La Tronche
  - CHRU Lille - Hôpital Claude Huriez, Clinique de Dermatologie, Lille
  - Hôpital La Timone, Marseille
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rouen-Hôpital, Rouen
  - Institut Gustave Roussy, Service de Dermatologie, Villejuif
- Germany (13):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Vivantes Klinikum Spandau, Dermatologie und Allergologie, Berlin
  - Universitaetsklinikum Koeln, Dermatologie und Venerologie,, Cologne
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Klinik und Poliklinik f. Dermatologie, Dresden
  - Helios Klinikum Erfurt, Dermatologie und Allergologie, Erfurt
  - Universitatsklinikum Essen Klinik fur Dermatologie Studienambulanz, Essen
  - Universitaetsklinikum Freiburg, Klinik fuer Dermatologie und Venerologie, Freiburg im Breisgau
  - Universitaetsklinikum Heidelberg, NCT-Dermatoonkologie, Heidelberg
  - Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Leipzig
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Hautklinik, Mainz
  - Universitaetsklinikum Mannheim, Klinik f. Dermatologie, Venerologie, Allergologle,, Mannheim
  - Studienzentrum Dermao-Onkologie, Universitaetsklinikum Tuebingen, Tübingen
- Italy (11):
  - Fondazione IRCCS CA'Granda Ospedale Maggiore Policlinico-Oncologia Medica, Milan, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano
  - A.O.S. Maria della Misericordia, Oncologia Medica, Perugia, Perugia
  - IRCCS Giovanni Paolo II Oncologia Medica, Bari
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Humanitas Istituto Clinico Catanese, U.O. Oncologia Medica, Misterbianco
  - Istituto Nazionale Tumori Fondazione G. Pascale, Oncologia Medica e Terapia Innovativa, Napoli
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone - U.O. Oncologia Medica, Palermo
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - A.O.U Senese Policlinico Santa Maria alle Scotte-UOC Immunoterapia Oncologica, Siena
  - Policlinico G.B. Rossi-Borgo Roma-Centro Ricerche Cliniche di Verona, Verona
- Japan (8):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Shinshu University Hospital, Matsumoto, Nagano
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - National Hospital Organization Osaka National Hospital, Chuo Ku, Osaka
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Nagaizumi-cho, Sunto-gun
  - The Cancer Institute Hospital of JFCR, Kōtoku, Tokho
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- Hospial Oncologico, Puerto Rico Medical Center, Rio Piedras, Puerto Rico, Puerto Rico
- National Cancer Centre, Singapore, Singapore
- South Africa (7):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Wilgers Oncology Centre, Pretoria, Gauteng
  - Curo Oncology, Pretoria, Gauteng
  - West Rand Oncology Centre Flora Clinic, Roodepoort, Gauteng
  - Excellentis Clinical Trial Consultants, George, Western Cape
  - Cape Town Oncology Trials Cape Gate Oncology Centre, Kraaifontein, Western Cape
  - Cancercare Rondebosch Oncology, Rondebosch, Western Cape
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Cha University Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Severance Hospital Younsei University Health System,, Seoul, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Chungnam National University Hospital, Daejeon, Jung-gu
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (12):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Catalan Institute of Oncology, Barcelona
  - ICO Badalona-Hospital Universitari Germans Trias I Pujol, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundación Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - Nuffield Health Wessex Hospital, Eastleigh, Hampshire
  - Edinburgh Cancer Center Western General Hospital, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MedlinePlus Genetics related topics: Melanoma — https://medlineplus.gov/genetics/condition/melanoma/
- See also: MedlinePlus related topics: Melanoma — https://medlineplus.gov/melanoma.html
- See also: Drug Information available for: Nivolumab — https://druginfo.nlm.nih.gov/drugportal/name/Nivolumab
- See also: Genetic and Rare Diseases Information Center resources: Neuroendocrine Tumor Neuroepithelioma — https://rarediseases.info.nih.gov/diseases/3963/neuroepithelioma
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks